CLINICAL TRIAL: NCT05776602
Title: Fast Brain MRI in Children With Suspected or Confirmed Brain Tumor
Brief Title: Fast Brain MRI in Children With Suspected Brain Tumor
Acronym: Fast MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anna Falk Delgado, MD, associate professor, Karolinska University Hospital
Other Study IDs: Fast Brain MRI in children
Record Dates: First submitted 2023-02-22; First posted 2023-03-20 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Magnetic Resonance Imaging; Brain Neoplasms, Childhood; Brain Neoplasms; Brain Tumor; Diagnosis; Image; Neuroimaging; Pediatric
Keywords: Neuro; Imaging; MRI; Diagnostic accuracy; Neuroimaging; Fast MRI; Neuromix; Pediatric
MeSH Terms: conditions — Brain Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients with suspected or confirmed brain tumor: New method och standard MRI in clinical care
  Interventions: Diagnostic Test: Fast MRI (Neuromix)

INTERVENTIONS:
Diagnostic Test: Fast MRI (Neuromix) — Diagnostic performance, correlation, agreement

SUMMARY:
This study aims to assess the diagnostic performance of a new fast MRI sequence named Neuromix compared to routine clinical MRI for brain tumor in pediatric patients

DETAILED DESCRIPTION:
The study aims to assess the diagnostic performance of fast MR sequence for the radiological evaluation of brain tumor in comparison to routine clinical MRI (or reference standard) in a pediatric population.

The primary outcome is the depiction and characterization of normal brain, brain tumor pathology and incidental findings.

Sensitivity, specificity, AUC and intra-/ interreader agreement for the diagnostic performance of Neuromix compared to cMRI will be obtained. Correlation of results between methods will be calculated.

Secondary outcomes will also include the assessment of diagnostic image quality and image artifacts.

The study population will consist of subjects aged 0-18 with a suspected or diagnosed brain tumor referred for routine MRI examination of the brain.

Study subjects will be investigated during the same day at 3T MR with Neuromix sequence in addition to the routine MRI examination.

Volume measurements will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18 years.
* Pediatric subjects with diagnosed or suspected brain tumor
* Referral routine MRI study.

Exclusion Criteria:

* MRI planned without sedation
* Aborted MR exam
* Unstable patient

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children up to 18 years with suspected or confirmed brain tumor investigated in standard clinical care with MRI of the brain.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | Through study completion, an average of 1 year
  AUC, area under the curve for the comparison of the new method against the reference standard

SECONDARY OUTCOMES:
Imaging artifacts | through study completion, an average of 1 year
  Image artifacts on both methods
Imaging quality | through study completion, an average of 1 year
  Image quality on both methods
Correlation | through study completion, an average of 1 year
  Correlation between readers and methods
Agreement | through study completion, an average of 1 year
  Agreement between readers and methods
Sensitivity | through study completion, an average of 1 year
  Sensitivity of the new method against the reference standard
Specificity | through study completion, an average of 1 year
  Specificity of the new method against the reference standard

CONTACTS AND LOCATIONS:
Overall Officials: Anna Falk Delgado, Ass Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinksa Universitetssjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No